CLINICAL TRIAL: NCT03367767
Title: Age-Related Eye Disease Study 2 (AREDS2) 10-Year Follow-On Study
Brief Title: Age-Related Eye Disease Study 2 (AREDS2) 10-year Follow-On
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 180023; 18-EI-0023
Record Dates: First submitted 2017-12-08; First posted 2017-12-11 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: AMD; Cancer; Cataract
Keywords: Blood Sample; Medical History; Optical Imaging
MeSH Terms: conditions — Neoplasms; Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Former AREDS2 and AREDS2 Follow-On participants

SUMMARY:
Background:

Age-related macular degeneration (AMD) and cataracts are two eye diseases. They were studied in the Age-Related Eye Disease Study (AREDS2) and the AREDS2 Follow-On study. These studies followed the natural course of the diseases. They also provided data on the long-term effects of certain oral supplements on AMD.

Objective:

To study the long-term effects of oral supplements on several things. These include incidences of lung cancer, development of late AMD, cataract surgery, cognitive function, and cardiovascular events.

Eligibility:

Former AREDS2 and AREDS2 Follow-On participants

Design:

Participants will have 1 visit. It will include:

An eye exam that tests how well participants can see, measures eye pressure, and checks eye movements. The pupil will be dilated with eye drops. Pictures will be taken of the retina and the inside of the eye.

Participants will grip a device in their hand to measure their grip strength.

A blood sample will be taken. This will be stored for future genetic research. Cells may be created from the sample.

A small sample of skin will be taken.

Sponsoring Institution: National Eye Institute

DETAILED DESCRIPTION:
Objective: The overall objective of this extended follow-up study is to provide data regarding the incidence of late age-related macular degeneration (AMD), cataract surgery and lung cancer in the approximately 1,200 AREDS2 study participants enrolled in the Follow-on study. The specific objectives for the study are to:

* Study the rates of progression to late AMD, neovascular AMD, or geographic atrophy associated with AMD.
* To seek incidences of lung cancer, by treatment assignment.
* To assess cognitive understanding by phone prior to coming into the clinic.
* To seek incidences of cardiovascular events.

Study Population: Up to 3,200 participants who were previously enrolled in the AREDS2 and AREDS2 Follow-on protocols are currently followed by telephone contact every six months for the past four years. It is expected that 1,200 of these 3,200 participants will be eligible to participate in the study. Up to 83 participants will be enrolled at the NEI.

Design: This is an extension of the multicenter, randomized trial of lutein, zeaxanthin and omega-3 polyunsaturated fatty acids in the AMD AREDS2 trial. Data for this extension will be collected by staff at selected AREDS2 clinical sites via an in-clinic visit.

Outcome Measures: The primary outcomes of the study will be the rates of progression to late AMD, neovascular AMD or geographic atrophy associated with AMD. Also of interest are the long-term rates of progression to late AMD, incidents of lung cancer and cataract surgery. Participant reports of incident cardiovascular events will be collected as secondary outcomes.

ELIGIBILITY:
* INCLUSION CRITERIA:

To participate in this study, the potential participant must meet all of the following criteria:

1. Previously enrolled in the AREDS2 and AREDS2 Follow-on protocols.
2. Participant must be offered sufficient opportunity to review and to understand the informed consent form, agree to the form s contents and provide written informed consent.

EXCLUSION CRITERIA:

There are no Exclusion Criteria.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Former AREDS2 and AREDS2 Follow-On participants
Sampling Method: Non-Probability Sample
Enrollment: 709 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
The incidence of advanced AMD, cataract surgery and lung cancer will be the primary outcomes of the study. | Study Completion

SECONDARY OUTCOMES:
Participant reports of incident cardiovascular events will be collected as secondary outcomes. | Study Completion

CONTACTS AND LOCATIONS:
Overall Officials: Emily Y Chew, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States